CLINICAL TRIAL: NCT00677677
Title: Safety and Immunogenicity of Human Papillomavirus (HPV) Vaccine in Solid Organ Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Assistant Professor of Medicine, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7350
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Transplant
Keywords: Lung transplant; Liver transplant; Kidney transplant; Pancreas transplant; HPV; Human Papillomavirus Quadrivalent Vaccine
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Human papillomavirus quadrivalent vaccine — Patients meeting the inclusion / exclusion criteria will be enrolled from outpatient transplant clinics. Upon enrolment, baseline serum will be obtained and patients will be given the first dose of vaccine. Two months later, serum will again be obtained and the second dose of vaccine will be administered. Finally, at month 6, serum will be obtained and the third dose of vaccine will be given. The final serum samples will be collected at months 7, 12 and 36. At 48 hours and 7 days after each vaccination, patients will be contacted by telephone for local and systemic adverse effect reporting.
  Other Names: Gardasil

SUMMARY:
Human papillomavirus (HPV) affects a significant number of transplant patients. In women, human papillomavirus (HPV) causes genital warts, pre-cancerous areas of the cervix, and cervical cancer. In men, the virus can cause warts of the anal and genital areas. Men can also sexually transmit the virus to their partners. A patient who has had an organ transplant is at higher risk of infections as well as cancers because of the lifelong immune suppressive medications. HPV vaccination is effective in the prevention of cervical cancer and is now recommended for all females aged 9-26 years by Alberta Health and Wellness and the Canadian National Advisory Committee on Immunization (NACI). However, how well the vaccine works in transplant patients is not known.

This study is being done to look at response of the immune system to HPV vaccine in men and women up to the age of 35 who have had an organ transplant. Men are also included in this study because they have the potential to get anal / genital warts and transmit the virus to their partners. The total duration of the study is three years. Fifty female and male solid organ transplant recipients (lung, heart, liver, kidney, pancreas, small bowel or combined organ transplants) on immunosuppression will be enrolled in the study.

DETAILED DESCRIPTION:
Cervical cancer affects a significant proportion of the female population. In Canada, it is estimated that there will be 1,350 new diagnoses of cervical cancer in 2007 and 390 deaths [1]. Human papillomavirus (HPV) is the causative agent in genital warts, cervical intraepithelial neoplasia, and cervical cancer. In this study, the vaccine will also be given to males, because males can develop anogenital warts and can transmit the virus to their partners. HPV is a nonenveloped DNA virus containing early and late genes. Although approximately 40 HPV types can infect the genital tract, only a few cause the majority of disease. For example, cancer-causing HPV includes HPV 16 whereas benign tumours are caused by HPV 6 [2].

HPV vaccine is a quadrivalent vaccine consisting of HPV types 6,11,16,18. Types 16 and 18 are implicated in the majority (~70%) of cervical cancers and at least half of CIN 2 and 3 lesions. Types 6 and 11 cause 90% of genital warts. The vaccine contains virus-like particles (VLPs) of the L1 proteins of the four serotypes and is adjuvanted with aluminum hydroxyphosphate sulphate. The vaccine does not contain live virions and cannot cause HPV disease. It is administered by intramuscular injection in three doses at 0, 2 months, and 6 months [2].

HPV vaccination is effective in the prevention of high grade cervical lesions and is now recommended for all females aged 9-26 years by the Canadian National Advisory Committee on Immunization (NACI) [3]. Although the vaccine is licensed for females, males can also develop anogenital warts and can transmit the virus to their partners. Immunogenicity trials have shown similar response to vaccine in adolescent males compared to females [15]. In addition, if women have been infected with 1-3 out of the four serotypes, vaccination appears to prevent cervical lesions from the remaining serotypes [16]. Therefore, although the vaccine is licensed for women ≤ 26 years old, it may also be applicable to somewhat older women who may not have acquired all four serotypes.

Solid organ transplantation is a life-saving modality; however, patients are on life-long immunosuppression which puts them at increased risk of infections as well as cancers. Studies have shown a high incidence of HPV infection in transplant recipients ranging from 17.5-45% [4-8]. An evaluation of 105 renal transplant recipients showed that 17.5% patients were infected with HPV [5]. Another study of 39 renal transplant recipients screened for HPV showed the presence of HPV in 30.7% of patients, primarily in the cervix [6]. Therefore, the risk of HPV infection has been estimated to be 17 times greater in renal transplant recipients than a matched immunocompetent population. Ano-genital neoplasia, related to HPV, is about 16-20 times more common in transplant recipients [5,6].

Yearly physical examinations of the anogenital area and annual Pap smears are recommended for transplant recipients [9]. However, there are no data on the immunogenicity of quadrivalent HPV vaccine in solid organ transplant recipients and no formal recommendations for vaccination in transplant recipients exist. Given that this is a patient population that is uniquely susceptible to HPV infection and its sequelae, it is important that vaccine immunogenicity be studied in transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Age ≥ 18 and ≤ 35
* Solid Organ Transplant ≥ 3 months post-transplant
* Outpatient status

Exclusion Criteria:

* Unable to comply with protocol
* Previous HPV vaccination
* Anticoagulation (that precludes intramuscular injection)
* Therapy for acute rejection in the past 2 weeks
* Febrile illness in the past 2 weeks
* Active CMV infection
* History of anogenital warts or cervical intraepithelial neoplasia or cervical cancer

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a 2-fold rise in the type-specific HPV titer for at least one of the four sertypes contained in the vaccine at month 7. | 36 months

SECONDARY OUTCOMES:
Vaccine adverse events including episodes of rejection up to 1 year after study enrolment. Immunogenicity at 36 months post-vaccination. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Barr E, Tamms G. Quadrivalent human papillomavirus vaccine. Clin Infect Dis. 2007 Sep 1;45(5):609-7. doi: 10.1086/520654. Epub 2007 Jul 25. PMID 17682997
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Human papillomavirus infection. Am J Transplant. 2004 Nov;4 Suppl 10:95-100. doi: 10.1111/j.1600-6135.2004.00732.x. No abstract available. PMID 15504222
- [Derived] Kumar D, Unger ER, Panicker G, Medvedev P, Wilson L, Humar A. Immunogenicity of quadrivalent human papillomavirus vaccine in organ transplant recipients. Am J Transplant. 2013 Sep;13(9):2411-7. doi: 10.1111/ajt.12329. Epub 2013 Jul 9. PMID 23837399